CLINICAL TRIAL: NCT03432390
Title: Continuous Positive Airway Pressure During General Anesthesia Induction For Elective Pediatric Surgery: Randomized Clinical Trial
Brief Title: Positive Pressure at Induction of Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Flavia orange, PhD, Clinical Professor, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 79591417.0.0000.5201
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Continuous Positive Airway Pressure; Hypoxia; General Anesthesia
MeSH Terms: conditions — Hypoxia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Experimental)
  Interventions: Device: Continuous Positive Airway Pressure
- Control (Active Comparator)
  Interventions: Device: Open system ventilation

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — A continuous positive airway pressure will be delivered to the patients during the induction of general anesthesia through the anesthesia work station
  Arms: CPAP
Device: Open system ventilation — Facemask ventilation adapted to the anesthesia work station
  Arms: Control

SUMMARY:
SCENARIO: Hypoxemia is one of the most common adverse events during the induction of general anesthesia and may culminate with more serious complications such as cardiac arrest and death. Pediatric patients, due to their anatomical and physiological characteristics, are more likely to develop hemoglobin desaturation levels. Some preventive strategies are used during this period to reduce the chances of occurrence of adverse event. Continuous Positive Airway Pressure (CPAP) may be useful during anesthetic induction in delaying the drop in oxygen levels in the blood by increasing this body gas reserves. OBJECTIVES: To assess the effectiveness of CPAP during anesthetic induction in increasing apnea time until hemoglobin saturation falls to 95% in children undergoing general anesthesia for elective surgery. METHODS: Phase III, parallel, randomized clinical trial to be developed at the Teaching Hospital of the Federal University of Pernambuco. Patients (72) are divided into two groups (36 in each) in which all patients will spontaneously ventilate: group C will receive CPAP and group A will use the open system. Children of pre-school age with physical status I or II, according to the American Anesthesia Society, candidates for elective surgery under general anesthesia will be included. Patients with pre-existing parenchymal lung disease, cyanotic children or patients with oxyhemoglobin saturation <95% prior to anesthetic induction and recent history (<4 weeks) or active upper respiratory tract infection will be excluded. The descriptive statistical analysis will be carried out through measures of central tendency and dispersion for quantitative variables and via distribution of frequencies for qualitative variables. ETHICAL ASPECTS: This work will respect human rights, principles of bioethics, the resolution 466/2012 of the National Health Council and the statement from Helsinki. Submission and approval by the research ethics committee is required prior to data collection. KEYWORDS: Continuous Positive Airway Pressure, Hypoxia, General Anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Pre-school children, ASA physical status I or II, Children undergoing general anesthesia for elective surgery

Exclusion Criteria:

* Pre-existing parenchymal lung disease, Children cyanotic or with oxyhemoglobin saturation less than 95% before anesthetic induction, Recent history (<4 weeks) or current upper respiratory tract infection

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arhem P, Klement G, Nilsson J. Mechanisms of anesthesia: towards integrating network, cellular, and molecular level modeling. Neuropsychopharmacology. 2003 Jul;28 Suppl 1:S40-7. doi: 10.1038/sj.npp.1300142. PMID 12827143
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Boonmak P, Boonmak S, Pattanittum P. High initial concentration versus low initial concentration sevoflurane for inhalational induction of anaesthesia. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD006837. doi: 10.1002/14651858.CD006837.pub2. PMID 22972100
- [Background] Park JH, Kim JY, Lee JM, Kim YH, Jeong HW, Kil HK. Manual vs. pressure-controlled facemask ventilation for anaesthetic induction in paralysed children: a randomised controlled trial. Acta Anaesthesiol Scand. 2016 Sep;60(8):1075-83. doi: 10.1111/aas.12737. Epub 2016 Apr 24. PMID 27109459
- [Background] von Ungern-Sternberg BS, Boda K, Chambers NA, Rebmann C, Johnson C, Sly PD, Habre W. Risk assessment for respiratory complications in paediatric anaesthesia: a prospective cohort study. Lancet. 2010 Sep 4;376(9743):773-83. doi: 10.1016/S0140-6736(10)61193-2. PMID 20816545
- [Background] Ehsan Z, Mahmoud M, Shott SR, Amin RS, Ishman SL. The effects of anesthesia and opioids on the upper airway: A systematic review. Laryngoscope. 2016 Jan;126(1):270-84. doi: 10.1002/lary.25399. Epub 2015 Jul 21. PMID 26198715
- [Background] Hedenstierna G, Edmark L. Effects of anesthesia on the respiratory system. Best Pract Res Clin Anaesthesiol. 2015 Sep;29(3):273-84. doi: 10.1016/j.bpa.2015.08.008. Epub 2015 Sep 18. PMID 26643094
- [Background] Bouroche G, Bourgain JL. Preoxygenation and general anesthesia: a review. Minerva Anestesiol. 2015 Aug;81(8):910-20. Epub 2015 Jun 5. PMID 26044934
- [Background] Nimmagadda U, Salem MR, Crystal GJ. Preoxygenation: Physiologic Basis, Benefits, and Potential Risks. Anesth Analg. 2017 Feb;124(2):507-517. doi: 10.1213/ANE.0000000000001589. PMID 28099321
- [Background] Gonzalez LP, Pignaton W, Kusano PS, Modolo NS, Braz JR, Braz LG. Anesthesia-related mortality in pediatric patients: a systematic review. Clinics (Sao Paulo). 2012;67(4):381-7. doi: 10.6061/clinics/2012(04)12. PMID 22522764
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Long E, Sabato S, Babl FE. Endotracheal intubation in the pediatric emergency department. Paediatr Anaesth. 2014 Dec;24(12):1204-11. doi: 10.1111/pan.12490. Epub 2014 Jul 15. PMID 25039321
- [Background] Bharti N, Batra YK, Kaur H. Paediatric perioperative cardiac arrest and its mortality: database of a 60-month period from a tertiary care paediatric centre. Eur J Anaesthesiol. 2009 Jun;26(6):490-5. doi: 10.1097/EJA.0b013e328323dac0. PMID 19300269
- [Background] Gonzalez LP, Braz JR, Modolo MP, de Carvalho LR, Modolo NS, Braz LG. Pediatric perioperative cardiac arrest and mortality: a study from a tertiary teaching hospital. Pediatr Crit Care Med. 2014 Nov;15(9):878-84. doi: 10.1097/PCC.0000000000000248. PMID 25226499
- [Background] Harless J, Ramaiah R, Bhananker SM. Pediatric airway management. Int J Crit Illn Inj Sci. 2014 Jan;4(1):65-70. doi: 10.4103/2229-5151.128015. PMID 24741500
- [Background] Chiron B, Mas C, Ferrandiere M, Bonnard C, Fusciardi J, Mercier C, Laffon M. Standard preoxygenation vs two techniques in children. Paediatr Anaesth. 2007 Oct;17(10):963-7. doi: 10.1111/j.1460-9592.2007.02259.x. PMID 17767632
- [Background] De Jong A, Futier E, Millot A, Coisel Y, Jung B, Chanques G, Baillard C, Jaber S. How to preoxygenate in operative room: healthy subjects and situations "at risk". Ann Fr Anesth Reanim. 2014 Jul-Aug;33(7-8):457-61. doi: 10.1016/j.annfar.2014.08.001. Epub 2014 Aug 29. PMID 25168301
- [Background] Humphreys S, Lee-Archer P, Reyne G, Long D, Williams T, Schibler A. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) in children: a randomized controlled trial. Br J Anaesth. 2017 Feb;118(2):232-238. doi: 10.1093/bja/aew401. PMID 28100527
- [Background] Windpassinger M, Plattner O, Gemeiner J, Roder G, Baumann A, Zimmerman NM, Sessler DI. Pharyngeal Oxygen Insufflation During AirTraq Laryngoscopy Slows Arterial Desaturation in Infants and Small Children. Anesth Analg. 2016 Apr;122(4):1153-7. doi: 10.1213/ANE.0000000000001189. PMID 26991620
- [Background] Faria DA, da Silva EM, Atallah AN, Vital FM. Noninvasive positive pressure ventilation for acute respiratory failure following upper abdominal surgery. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD009134. doi: 10.1002/14651858.CD009134.pub2. PMID 26436599
- [Background] Bratton DJ, Stradling JR, Barbe F, Kohler M. Effect of CPAP on blood pressure in patients with minimally symptomatic obstructive sleep apnoea: a meta-analysis using individual patient data from four randomised controlled trials. Thorax. 2014 Dec;69(12):1128-35. doi: 10.1136/thoraxjnl-2013-204993. Epub 2014 Jun 19. PMID 24947425
- [Background] Wang J, Yu W, Gao M, Zhang F, Li Q, Gu C, Yu Y, Wei Y. Continuous positive airway pressure treatment reduces cardiovascular death and non-fatal cardiovascular events in patients with obstructive sleep apnea: A meta-analysis of 11 studies. Int J Cardiol. 2015 Jul 15;191:128-31. doi: 10.1016/j.ijcard.2015.05.003. Epub 2015 May 5. No abstract available. PMID 25965619
- [Background] Iftikhar IH, Khan MF, Das A, Magalang UJ. Meta-analysis: continuous positive airway pressure improves insulin resistance in patients with sleep apnea without diabetes. Ann Am Thorac Soc. 2013 Apr;10(2):115-20. doi: 10.1513/AnnalsATS.201209-081OC. PMID 23607839
- [Background] de Freitas Dantas Gomes EL, Costa D, Germano SM, Borges PV, Sampaio LM. Effects of CPAP on clinical variables and autonomic modulation in children during an asthma attack. Respir Physiol Neurobiol. 2013 Aug 1;188(1):66-70. doi: 10.1016/j.resp.2013.05.004. Epub 2013 May 13. PMID 23681081
- [Background] Jat KR, Mathew JL. Continuous positive airway pressure (CPAP) for acute bronchiolitis in children. Cochrane Database Syst Rev. 2015 Jan 7;1:CD010473. doi: 10.1002/14651858.CD010473.pub2. PMID 25563827
- [Background] Sinha IP, McBride AKS, Smith R, Fernandes RM. CPAP and High-Flow Nasal Cannula Oxygen in Bronchiolitis. Chest. 2015 Sep;148(3):810-823. doi: 10.1378/chest.14-1589. PMID 25836649
- [Background] Wilson PT, Morris MC, Biagas KV, Otupiri E, Moresky RT. A randomized clinical trial evaluating nasal continuous positive airway pressure for acute respiratory distress in a developing country. J Pediatr. 2013 May;162(5):988-92. doi: 10.1016/j.jpeds.2012.10.022. Epub 2012 Nov 16. PMID 23164308
- [Background] Sreejit MS, Ramkumar V. Effect of positive airway pressure during pre-oxygenation and induction of anaesthesia upon safe duration of apnoea. Indian J Anaesth. 2015 Apr;59(4):216-21. doi: 10.4103/0019-5049.154998. PMID 25937647
- [Background] Harbut P, Gozdzik W, Stjernfalt E, Marsk R, Hesselvik JF. Continuous positive airway pressure/pressure support pre-oxygenation of morbidly obese patients. Acta Anaesthesiol Scand. 2014 Jul;58(6):675-80. doi: 10.1111/aas.12317. Epub 2014 Apr 16. PMID 24738713
- [Background] Squadrone V, Coha M, Cerutti E, Schellino MM, Biolino P, Occella P, Belloni G, Vilianis G, Fiore G, Cavallo F, Ranieri VM; Piedmont Intensive Care Units Network (PICUN). Continuous positive airway pressure for treatment of postoperative hypoxemia: a randomized controlled trial. JAMA. 2005 Feb 2;293(5):589-95. doi: 10.1001/jama.293.5.589. PMID 15687314
- [Background] Pradhapan P, Swaminathan M, Salila Vijayalal Mohan HK, Sriraam N. Identification of apnea during respiratory monitoring using support vector machine classifier: a pilot study. J Clin Monit Comput. 2013 Apr;27(2):179-85. doi: 10.1007/s10877-012-9411-8. Epub 2012 Nov 21. PMID 23179018
- [Background] Simon BA, Kaczka DW, Bankier AA, Parraga G. What can computed tomography and magnetic resonance imaging tell us about ventilation? J Appl Physiol (1985). 2012 Aug 15;113(4):647-57. doi: 10.1152/japplphysiol.00353.2012. Epub 2012 May 31. PMID 22653989
- [Background] Jubran A. Pulse oximetry. Crit Care. 2015 Jul 16;19(1):272. doi: 10.1186/s13054-015-0984-8. PMID 26179876
- [Background] Roy WL, Lerman J. Laryngospasm in paediatric anaesthesia. Can J Anaesth. 1988 Jan;35(1):93-8. doi: 10.1007/BF03010554. No abstract available. PMID 3280151
- [Background] Pitrez PM, Pitrez JL. [Acute upper respiratory tract infections: outpatient diagnosis and treatment]. J Pediatr (Rio J). 2003 May;79 Suppl 1:S77-86. doi: 10.2223/jped.1002. Portuguese. PMID 14506520
- [Background] Saklad M. Grading of patients for surgical procedures. Anesthesiology. 1941;2(3):281-284
- [Background] ASA Physical Status Classification System. https://www.asahq.org/resources/clinical-information/asa-physical-status-classification-system. Published 2014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the Teaching Hospital of the Federal University of Pernambuco
Pre-assignment Details: Ninety-eight patients were screened for the purpose of determining eligibility; seventy-two were enrolled, twenty-six were not due to not meeting the inclusion criteria [ASA >2,(01); Not Preschool-aged (21)], meeting the exclusion criteria [current upper respiratory tract infection(03)] or not signing the written informed consent (01)
Groups:
- Control: Open System Ventilation: Open system ventilation: Facemask ventilation adapted to the anesthesia work station
Period: Apnea Period
Arm/Group | CPAP | Control: Open System Ventilation
Started | 36 | 36
Completed | 34 | 34
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 2
Period: Recovery Period
Arm/Group | CPAP | Control: Open System Ventilation
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP | Control: Open System Ventilation | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.34 (1.44) | 4.23 (1.51) | 4.28 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 28 | 24 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 34 | 34 | 68
American Society of Anesthesiologists Physical Status [Count of Participants; unit: Participants] — State based on the presence / absence of disease in the patients or on non-pathological physiological changes, as well as the quality of the control of morbidities. Ordinal variable whose categories are numbered in digits I to VI, with states I, absence of systemic disease, and II, systemic disease controlled
  Participants
    Physical Status I | 31 | 33 | 64
    Physical Status II | 3 | 1 | 4
Weight [Mean (Standard Deviation); unit: kilograms] | 18.28 (4.87) | 17.77 (4.58) | 18.03 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Time Between Onset of Apnea and the Drop in 95% Oxyhemoglobin Saturation Levels
Description: In children undergoing general anesthesia for elective surgery who will undergo CPAP or standard circular circuit ventilation during anesthesia induction, compare the time between onset of apnea and the drop in 95% oxyhemoglobin saturation between the groups
Time Frame: During induction of general anesthesia (up to five minutes after beginning of apnea)
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- Controle: Open system ventilation: Facemask ventilation adapted to the anesthesia work station
Arm/Group | CPAP | Controle
Number analyzed (Participants) | 34 | 34
seconds | 227.65 [198.08 to 257.21] | 133.68 [109.11 to 158.24]
Statistical Analysis 1: Comparison: CPAP vs Controle; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Time to Recovery of Oxyhemoglobin Saturation Levels in Pre-apnea Pulse Oximetry
Description: In children undergoing general anesthesia for elective surgery who will undergo CPAP or standard circular circuit ventilation during anesthesia induction, compare: The time to recovery of oxyhemoglobin saturation levels in pre-apnea pulse oximetry between groups
Time Frame: During induction of general anesthesia (up to five minutes after beginning of apnea)
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | CPAP | Controle
Number analyzed (Participants) | 34 | 34
Seconds | 38.65 [13.42 to 63.87] | 43.12 [21.26 to 64.99]

3. Secondary Outcome: Number of Participants That Experienced Complications While Undergoing General Anesthesia
Description: In children undergoing general anesthesia for elective surgery who will undergo CPAP or standard circular circuit ventilation during anesthesia induction, compare: The frequency of complications (laryngospasm, hypoxemia, bradycardia, cardiorespiratory arrest, death) between the groups
Time Frame: During induction of general anesthesia (up to five minutes after beginning of apnea)
Measure: Count of Participants; unit: Participants
Arm/Group | CPAP | Controle
Number analyzed (Participants) | 34 | 34
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Five minutes
Arm/Group | CPAP | Control: Open System Ventilation
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT03432390/Prot_SAP_ICF_000.pdf